CLINICAL TRIAL: NCT03691012
Title: Circulating Tumour DNA as a Marker of Residual Disease and Response to Adjuvant Chemotherapy in Stage I-IV Epithelial Ovarian, Fallopian Tube and Primary Peritoneal Cancer (EOC)
Brief Title: Circulating Tumour DNA as a Marker of Residual Disease & Response to Adjuvant Chemotherapy in Stage I-IV Ovarian Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Walter and Eliza Hall Institute of Medical Research (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Maria Edmonds, Assoc Professor Sumitra Ananda, Walter and Eliza Hall Institute of Medical Research
Other Study IDs: WEHI-ctDNA-10
Record Dates: First submitted 2018-03-11; First posted 2018-10-01 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Using the Safe-SeqS assay, the fraction of total DNA fragments (mutant and wild-type) of a given gene that contains the queried mutation will be determined. In cases where mutations are acquired in the tumour, mutant DNA fragments are expected to represent only a small fraction of the total DNA fragments in the circulation. In cases with germline BRCA mutations, where normal or non-tumour cells also harbour the specific DNA changes, we would expect to find the fraction of mutant DNA for a given gene to be much higher. If unexpected results are found for mutations, indicating the possibility of an inherited mutation, the patient will be informed of the result by their treating doctor and the potential implication.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Circulating tumour DNA testing — Circulating tumour DNA testing

SUMMARY:
To demonstrate that detectable ctDNA in peripheral blood following debulking of the primary tumour or following completion of adjuvant treatment for is associated with subsequent disease recurrence in stage I-IV epithelial, fallopian tube and primary peritoneal cancer (Ovarian Cancer)

DETAILED DESCRIPTION:
This is a prospective,multi-centre study involving serial blood collections from 100 stage I-IV debulked (or to be debulked in the case of neoadjuvant chemotherapy) high grade serous, endometrioid and clear cell ovarian, fallopian tube and primary peritoneal cancer patients (EOC) or ovarian carcinosarcoma planned to receive adjuvant chemotherapy. Tumour samples will be made available following patient enrollment for the primary debulking group, and following surgery for the neoadjuvant group for mutation analysis. Ascites will not be accepted. Up to four blood samples in the primary debulking group and up to five blood samples in the neoadjuvant group will be collected from each patient over a 6-8 month period for ctDNA and Ca125 analysis Choice of chemotherapy will be platinum based treatment at the treating clinician's discretion as per standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Patients that have had primary debulking surgery for curatively resected stage I-IV high grade serous, endometrioid or clear cell carcinoma, or carcinosarcoma of the ovary, fallopian tube or primary peritoneum. Stage IV patients can only be included in the study if they have had a complete resection of all macroscopic disease with no residual disease.

   OR Patients commencing neoadjuvant chemotherapy for stage I- III high grade serous, endometrioid or clear cell carcinoma, or carcinosarcoma of the ovary, fallopian tube or primary peritoneum. Women must be planned to undergo interim debulking surgery.
2. A representative tumour sample can be made available for molecular testing after surgery or a core biopsy pre neoadjuvant chemotherapy if available.
3. Fit and planned for adjuvant chemotherapy

Exclusion Criteria:

1. History of another primary cancer within the last 3 years
2. Patients with Epithelial Ovarian, Fallopian Tube and Primary Peritoneal Cancer (EOC) of mucinous subtype and sarcoma
3. Patients with Stage IV disease who have residual disease
4. Patients <18 years

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Ovarian Cancer
Study Population: Patients that have had primary debulking surgery for curatively resected stage I-IV high grade serous, endometrioid or clear cell carcinoma, or carcinosarcoma of the ovary, fallopian tube or primary peritoneum. Stage IV patients can only be included in the study if they have had a complete resection of all macroscopic disease with no residual disease.OR Patients commencing neoadjuvant chemotherapy for stage I- III high grade serous, endometrioid or clear cell carcinoma, or carcinosarcoma of the ovary, fallopian tube or primary peritoneum. Women must be planned to undergo interim debulking surgery.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2025-05-09 (Estimated)

PRIMARY OUTCOMES:
Circulating DNA in the plasma of cancer patients has been shown to exhibit tumour-related alteration. These mutations in tumour cells,can be used as highly specific biomarkers of disease burden. Baseline. | After surgery (primary debulking group) or pre cycle 1 of therapy (neoadjuvant) confirmed with conventional radiological imaging and CA125 (cycles of chemotherapy are 21 days in length).
  polymerase chain reaction (PCR) to quantify ctDNA

SECONDARY OUTCOMES:
Circulating DNA in the plasma of cancer patients has been shown to exhibit tumour-related alteration. These mutations in tumour cells can be used as highly specific biomarkers of disease burden. Change from baseline and previous result. | At the completion of pre cycle 3 of chemotherapy (primary debulking group) confirmed with Convential Radiological imaging and CA125. (each cycle 21 days in length)
  polymerase chain reaction (PCR) to quantify ctDNA
Circulating DNA in the plasma of cancer patients has been shown to exhibit tumour-related alteration. These mutations in tumour cells can be used as highly specific biomarkers of disease burden. Change from baseline and previous result. | circulating tumour DNA (ctDNA) during chemotherapy pre cycle 5 confirmed (primary debluking group) with conventional Radiological imaging and CA125 (each cycle 21 days in length).
  polymerase chain reaction (PCR) to quantify ctDNA
Circulating DNA in the plasma of cancer patients has been shown to exhibit tumour-related alteration. These mutations in tumour cells can be used as highly specific biomarkers of disease burden. Change from baseline and previous result | circulating tumour DNA (ctDNA) during chemotherapy pre cycle 3 or 4 (neoadjuvant group) confirmed with conventional Radiological imaging and CA125 (each cycle 21 days in length)
  polymerase chain reaction (PCR) to quantify ctDNA
Circulating DNA in the plasma of cancer patients has been shown to exhibit tumour-related alteration. These mutations in tumour cells can be used as highly specific biomarkers of disease burden. Change from baseline and previous result. | At the completion of 6 of chemotherapy (primary debulking group) confirmed with conventional Radiological imaging and CA125 (each cycle 21 days in length)
  polymerase chain reaction (PCR) to quantify ctDNA
Circulating DNA in the plasma of cancer patients has been shown to exhibit tumour-related alteration. These mutations in tumour cells can be used as highly specific biomarkers of disease burden. Change from baseline and previous result. | At the completion of 6 cycles of chemotherapy (neoadjuvant group) confirmed with conventional radiology and CA125 (at the end of 18 weeks).
  polymerase chain reaction (PCR) to quantify ctDNA

CONTACTS AND LOCATIONS:
Overall Officials: Sumitra Ananda, Associate Professor, Principal Investigator — Walter and ELiza Hall Institute
Locations (7):
- John Hopkins University School of Medicine, Baltimore, Maryland, United States
- Australia (6):
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Epworth Freemasons, Melbourne, Victoria
  - Western Hospital, Melbourne, Victoria
  - Mercy Hospital for Women, Melbourne, Victoria
  - Cabrini Malvern, Melbourne, Victoria
  - Monash Medical Centre, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No
All patients will be provided with a unique code number for the purposes of transferring information. Any data that leave the hospital will be coded. this information does not include patient's name or other personal identifiers